CLINICAL TRIAL: NCT05722236
Title: A Randomized, Wait List-Controlled, Clinical Trial of IBD Strong Peer for Self-Management of Psychological Distress by Persons Living With Inflammatory Bowel Diseases (IBD)
Brief Title: IBD Strong Peer2Peer for Self-Management of Psychological Distress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Jones (Other)
Collaborators: Crohn's and Colitis Canada (Other); Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Jennifer Jones, Clinical Gastroenterologist, Associate Professor, Department of Medicine, Dalhousie University, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 50596
Record Dates: First submitted 2022-12-22; First posted 2023-02-10 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
Keywords: peer mentoring; psychological distress; IBD; mental health; access
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IBD Strong Peer2Peer intervention (Experimental)
  Interventions: Behavioral: IBD Strong Peer2Peer
- Waitlist -controls (Other)
  Interventions: Other: Waitlist control

INTERVENTIONS:
Behavioral: IBD Strong Peer2Peer — Mentee participants will experience the intervention: this group will partake in peer-led sessions (peer calls) consisting of up to 10 virtual sessions on Zoom lasting approximately 20-30 minutes in duration over eight weeks. Individual peer calls will be unstructured whereby trained mentors (patients with IBD who have undergone training to be a mentor) and mentees will be given the freedom to discuss whatever issues they choose. Psychological and emotional support is provided to the mentee by the mentor.
  Arms: IBD Strong Peer2Peer intervention
Other: Waitlist control — Wait list controls will be offered participation in the IBD Strong Peer2Peer intervention once post-control outcome measures have been completed.
  Arms: Waitlist -controls

SUMMARY:
Psychological distress (PD) as a result of inflammatory bowel disease (IBD) is prevalent and associated with worse disease-related outcomes. IBD-associated psychological distress (IBD-PD) is particularly common at initial diagnosis, during disease flares, before surgery, and during transitions of care. Access to evidence-based, gold-standard psychological interventions and emotional support for IBD-PD has been identified as a major care gap by persons living with IBD. The COVID-19 pandemic has further exacerbated the burden of PD for persons living with chronic diseases like IBD, predisposing at-risk individuals to even greater mental struggles. Studies have shown a minority of patients are asked about IBD-PD in routine clinical care and that even if asked, access to mental health care is extremely limited. iPeer2Peer is an evidence-based, peer-led, virtually administered intervention for IBD-PD in the pediatric population that has demonstrated feasibility, acceptability and early effectiveness. Using qualitative data derived from an extensive stakeholder engagement process, iPeer2Peer has been adapted to meet the needs of adults living with IBD-PD. This program, IBD Strong Peer, will be studied through a randomized, wait list-controlled hybrid implementation-effectiveness trial in Nova Scotia. This study will provide implementation data needed to improve and adapt the intervention and implementation strategy to meet local needs, as well as provide early effectiveness data. This data will inform the design and statistical power needed for future larger, multicenter randomized control trials. IBD Strong Peer has significant potential to improve access to evidence-informed interventions for IBD-PD.

ELIGIBILITY:
Inclusion Criteria:

* Adult IBD patient (18 years or older)
* In a period of transition (newly diagnosed, transitioning from pediatric to adult care, flaring or changing medications, recently admitted to hospital, or facing the need for surgery)

Exclusion Criteria:

* Screening positive for severe psychological pathology
* Do not speak English
* Diagnosis of a major comorbid psychiatric condition such as bipolar disorder or schizophrenia,
* No access to the internet

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Participant Satisfaction | week 4
  Satisfaction, measured by the satisfaction questionnaire: QUOTE IBD, where QI index < 0.9 = suboptimal satisfaction)
Participant Satisfaction | week 8
  Satisfaction, measured by the satisfaction questionnaire: QUOTE IBD, where QI index < 0.9 = suboptimal satisfaction)
Attrition rate | week 4
  Rate of participants who drop out of the study
Attrition rate | week 8
  Rate of participants who drop out of the study
Adherence rate | week 4
  Rate of participants who adhere to the study protocol
Adherence rate | week 8
  Rate of participants who adhere to the study protocol
Recruitment success | Pre-study Baseline
  recruitment success [participation/ total number approached or referred]
Recruitment success | week 4
  recruitment success [participation/ total number approached or referred]
Recruitment success | week 8
  recruitment success [participation/ total number approached or referred]
Fidelity | week 1
  Audio recording of session to determine what interventions were delivered, intervention fidelity (Module content completion will be assessed via thematic analysis).
Fidelity | week 2
  Audio recording of session to determine what interventions were delivered, intervention fidelity (Module content completion will be assessed via thematic analysis).
Fidelity | week 3
  Audio recording of session to determine what interventions were delivered, intervention fidelity (Module content completion will be assessed via thematic analysis).
Fidelity | week 4
  Audio recording of session to determine what interventions were delivered, intervention fidelity (Module content completion will be assessed via thematic analysis).
Fidelity | week 5
  Audio recording of session to determine what interventions were delivered, intervention fidelity (Module content completion will be assessed via thematic analysis).
Fidelity | week 6
  Audio recording of session to determine what interventions were delivered, intervention fidelity (Module content completion will be assessed via thematic analysis).
Fidelity | week 7
  Audio recording of session to determine what interventions were delivered, intervention fidelity (Module content completion will be assessed via thematic analysis).
Fidelity | week 8
  Audio recording of session to determine what interventions were delivered, intervention fidelity (Module content completion will be assessed via thematic analysis).
General quality of life score (Eq5D-3L ) | Pre-study Baseline
  General quality of life score measured by the European Quality of Life 5 Dimensions 3 Level Version (Eq5D-3L) index
General quality of life score (Eq5D-3L ) | week 4
  General quality of life score measured by the European Quality of Life 5 Dimensions 3 Level Version (Eq5D-3L) index
General quality of life score (Eq5D-3L ) | week 8
  General quality of life score measured by the European Quality of Life 5 Dimensions 3 Level Version (Eq5D-3L) index
General quality of life score (SF-36) | Pre-study baseline
  General quality of life score measured by the SF-36 questionnaire
General quality of life score (SF-36) | week 4
  General quality of life score measured by the SF-36 questionnaire
General quality of life score (SF-36) | week 8
  General quality of life score measured by the SF-36 questionnaire
IBD Related quality of life score | Pre-study baseline
  IBD Related quality of life score, measured by the Short Inflammatory Bowel Disease Questionnaire (SIBDQ)
IBD Related quality of life score | week 4
  IBD Related quality of life score, measured by the Short Inflammatory Bowel Disease Questionnaire (SIBDQ)
IBD Related quality of life score | week 8
  IBD Related quality of life score, measured by the Short Inflammatory Bowel Disease Questionnaire (SIBDQ)
Participant Self efficacy score | Pre-study Baseline
  Self-efficacy, measured by the New General Self Efficacy Scale
Participant Self efficacy score | week 4
  Self-efficacy, measured by the New General Self Efficacy Scale
Participant Self efficacy score | week 8
  Self-efficacy, measured by the New General Self Efficacy Scale
Psychological distress (DSM-V) | Pre-study Baseline, week 4 and week 8
  Participant psychological distress, measured by the DSM-V cross cutting questionnaire
Psychological distress (DSM-V) | week 4
  Participant psychological distress, measured by the DSM-V cross cutting questionnaire
Psychological distress (DSM-V) | week 8
  Participant psychological distress, measured by the DSM-V cross cutting questionnaire
Psychological distress (PSS) | Pre-study Baseline
  Participant psychological distress, measured by the Perceived Stress Scale (PSS)
Psychological distress (PSS) | week 4
  Participant psychological distress, measured by the Perceived Stress Scale (PSS)
Psychological distress (PSS) | week 8
  Participant psychological distress, measured by the Perceived Stress Scale (PSS)
Psychological distress (GAD7) | Pre-study Baseline
  Participant psychological distress, measured by the Generalized Anxiety Disorder Assessment (GAD7) scale
Psychological distress (GAD7) | week 4
  Participant psychological distress, measured by the Generalized Anxiety Disorder Assessment (GAD7) scale
Psychological distress (GAD7) | week 8
  Participant psychological distress, measured by the Generalized Anxiety Disorder Assessment (GAD7) scale
Psychological distress (PHQ8) | Pre-study Baseline
  Participant psychological distress, measured by the eight-item Patient Health Questionnaire depression (PHQ8) scale
Psychological distress (PHQ8) | week 4
  Participant psychological distress, measured by the eight-item Patient Health Questionnaire depression (PHQ8) scale
Psychological distress (PHQ8) | week 8
  Participant psychological distress, measured by the eight-item Patient Health Questionnaire depression (PHQ8) scale

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre, Halifax, N.S., Canada

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391